CLINICAL TRIAL: NCT03618836
Title: Study of the Risk of PREMaturité According to the Balance of Bacterial Flora VAginale (PREMEVA2)
Brief Title: Study of the Risk of PREMaturité According to the Balance of Bacterial Flora VAginale
Acronym: PREMEVA2
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011_16; 2011-A01254-37 (Other: ID-RCB number, ANSM); PHRC_N 2011N°19-22 (Other: PHRC number)
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Preterm Birth
Keywords: Bacterial vaginosis; Vaginal microbiota; Molecular methods; Next generation sequencing
MeSH Terms: conditions — Premature Birth; Vaginosis, Bacterial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal samples with DNA of microorganisms
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases. Preterm Births: Microbiological and biological patterns on vaginal samples in the first trimester of pregnancy among spontaneous preterm births between 22 and 36 weeks
  Interventions: Other: Microbiological and biological patterns on vaginal samples
- Controls. Term Births: Microbiological and biological patterns on vaginal samples in the first trimester of pregnancy among deliveries over ≥ 37 weeks
  Interventions: Other: Microbiological and biological patterns on vaginal samples

INTERVENTIONS:
Other: Microbiological and biological patterns on vaginal samples — To compare the microbiological and biological patterns between groups

SUMMARY:
Objective

To compare vaginal microbiota in the first trimester of pregnancy between spontaneous preterm and term deliveries

DETAILED DESCRIPTION:
Material and methods Case-control study nested in a cohort of pregnant patients in the first trimester. Inclusion criteria. : case is defined as spontaneous preterm births between 22 and 36 weeks in one of the 14 centers. The "control" patient will be considered as the following delivery over ≥ 37 weeks in the same center.

Multiple pregnancies, medical interruptions of pregnancy and deaths in utero will be excluded. Regarding the vaginal flora of cases and controls, the microorganisms will be researched and quantified by molecular methods.

Expected results

Patients and control patients will be compared for their demographic, obstetric, clinical and microbiological data. The parameters related to the risk of spontaneous prematurity at the p <0.20 threshold will then be analyzed by multi-level logistic regression.

Implications At a time when the link between bacterial vaginosis and prematurity is controversial, the detection - or not - of microorganisms linked to the risk of prematurity will be a key issue.

ELIGIBILITY:
Inclusion Criteria:

* case: spontaneous preterm births between 22 and 36 weeks in one of the 14 centers
* controls : the following delivery over ≥ 37 weeks in the same center

Exclusion Criteria:

* Multiple pregnancies, medical interruptions of pregnancy and deaths in utero

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Cohort of pregnant patients in the first trimester
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Vaginal Microbiota pattern | 10 years
  All microorganism potentially present in the vagina

SECONDARY OUTCOMES:
Vaginal biological pattern | 10 years
  Biochemical and immunological compounds present in the vagina

CONTACTS AND LOCATIONS:
Overall Officials: Damien Subtil, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No